CLINICAL TRIAL: NCT07106931
Title: Early STratification of Acute ARThritis (START)- A Prospective Observational Study
Brief Title: Early STratification of Acute ARThritis
Acronym: START
Status: Recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Silje Watterdal Syversen, MD PhD, Diakonhjemmet Hospital
Other Study IDs: REC671173
Record Dates: First submitted 2025-06-03; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Arthritis
Keywords: early onset arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, synovial fluid and synovial biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational study with no intervention — This is an observational study with no intervention

SUMMARY:
The prospective observational study "Early STratification of acute inflammatory ARThritis" (START) aims to build a platform for identification of markers for early stratification of inflammatory arthritis to ensure timely diagnosis and correct initial treatment. Management of early-stage inflammatory arthritis is a daily challenge for the rheumatologist and encompasses a range of conditions. Stratification is needed both for optimal diagnostics and for personalising therapy, but is hampered by a lack of tools. Current evaluation is inadequate for early diagnosis and treatment of inflammatory joint diseases as well as for timely diagnosis of infections. The clinical role of novel biomarkers needs to be investigated in large patient samples. In the START study, an extensive data collection will be performed to build a platform for identification and validation of biomarkers for stratification of early-stage inflammatory arthritis. The study has an ambitious goal of improving patient care by increased understanding of the disease. The project applies a unique multitude of approaches to characterisation of patients, including modern imaging techniques, analyses of synovial fluid and -biopsies, genetic and epigenetic markers, proteomics, microbiota analyses and immunological markers. The results will enable clinicians to make better informed treatment decisions for the individual patient with early-stage inflammatory arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Arthritis* in one or more joints of less than 12 weeks' duration**
* Adult patients (> 18 years) capable of understanding and signing an informed consent form

  * Defined as currently active clinical synovitis (ie, swelling) in at least one joint as determined by an expert assessor which might be confirmed by ultrasonography ** Prior patient reported swollen joint not confirmed as arthritis by a rheumatologist is not an exclusion

Exclusion Criteria:

* Swollen joint related to trauma
* Subject not capable of adhering to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients refered to the outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2044-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
Final diagnosis | 12 months
  Number of patients with a final diagnoses of the differnent forms of arthritis assed by the ICD-10 codes given by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet